CLINICAL TRIAL: NCT02305160
Title: Phase 3 Multicenter, Randomized, Open Label Trial of a New Low Cost Animal Extracted Surfactant to Treat Respiratory Distress Syndrome in Preterm Infants
Brief Title: A Multicenter, Randomized, Open Label Trial of a New Animal Extracted Surfactant to Treat RDS in Preterm Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Celso Moura Rebello, MD PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012005B
Record Dates: First submitted 2014-02-26; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory distress syndrome; Pulmonary surfactant; Mortality; Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — beractant; poractant alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Butantan (Experimental): The new pulmonary surfactant produced by Butantan Institute. Butantan Surfactant: 100 mg/kg, IT, maximum of 3 doses.
  Interventions: Drug: Butantan
- Control (Active Comparator): The pulmonary surfactants commercially available in Brazil Survanta or Curosurf: 100 mg/kg, IT, maximum of 3 doses.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Butantan — Use of Butantan surfactant 100 mg/kg, IT, maximum of 3 doses
  Other Names: Butantan Surfactant
  Arms: Butantan
Drug: Control — The pulmonary surfactants commercially available in Brazil Survanta or Curosurf: 100 mg/kg, IT, maximum of 3 doses.
  Other Names: Survanta or Curosurf
  Arms: Control

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the new pulmonary surfactant produced by Butantan Institute among premature infants with gestational age below 34 weeks with RDS, comparing to the pulmonary surfactants commercially available in Brazil.

DETAILED DESCRIPTION:
Exogenous surfactant replacement therapy has been one of the major advances in the treatment of premature infants with respiratory distress syndrome (RDS). It has decreased the mortality among premature infants with RDS, determining changes in the children mortality rates among the developed countries. High cost, however, has been a major handicap for its wide use in developing and underdeveloped countries. Based on that, Butantan Institute (Sao Paulo, Brazil) has developed a new porcine pulmonary surfactant preparation at lower production cost. Initial animal studies showed similar improvement in lung mechanics and histopathologic findings to those observed with commercially available preparations.

Comparison(s): The new surfactant developed and produced by Butantan Institute will be compared to the commercially available pulmonary surfactants in Brazil, regarding to the efficiency to maintain a good arterial oxygenation, low airway pressures after treatment, similar mortality rates, and similar rates of complications like bronchopulmonary dysplasia and pulmonary hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age below 34 weeks
* RDS diagnosis based on clinical and RDS radiographic patterns
* Need of mechanical ventilation
* Parental consent

Exclusion Criteria:

* Age greater than 24 hours
* Major congenital malformations
* Unstable hemodynamic status
* Occurence of seizure during the stay in the Neonatal Intensive Care Unit
* Maternal and/or fetal infection (chorioamnionitis: maternal fever, foul vaginal discharge, fetal tachycardia, uterine tenderness, leukocytosis or leukopenia) or congenital infection

Ages: 1 Minute to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 327 (Actual)
Dates: Start 2005-04; Primary Completion 2006-05 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 72 hours after treatment
  Mortality rate 72 hours after treatment

SECONDARY OUTCOMES:
The incidence of adverse effects as: pneumothorax, pneumomediastinum, pulmonary interstitial emphysema, pulmonary hemorrhage and bronchopulmonary dysplasia (BPD). | 28 days of life
  Incidence of main complications of prematurity at 28 days of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Precioso, MD PhD, Study Director — University of Sao Paulo Medical School Department of Pediatrics; Celso M Rebello, MD PhD, Principal Investigator — University of Sao Paulo Medical School - Department of Pediatrics; Renata S Mascaretti, MD PhD, Study Director — University of Sao Paulo Medical School Department of Pediatrics
Locations (30):
- Brazil (30):
  - Hospital Esau de Matos, Vitória da Conquista, Estado de Bahia
  - Hospital Regional de Taguatinga, Brasília, Federal District
  - Hospital Materno Infantil, Goiânia, Goiás
  - Hospital Universitario - Unidade Materno Infantil, São Luís, Maranhão
  - Maternidade Odete Valadares, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de BH, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Sofia feldman, Belo Horizonte, Minas Gerais
  - Hospital Municipal Odilon Behrens, Belo Horizonte, Minas Gerais
  - Hospital Julia Kubstchek, Belo Horizonte, Minas Gerais
  - IMIP, Recife, Pernambuco
  - Hospital Barao de Lucena, Recife, Pernambuco
  - CISAM - Universidade de Pernambuco, Recife, Pernambuco
  - Hospital Maternidade Oswaldo de Nazareth, Rio de Janeiro, Rio de Janeiro
  - Hospital Maternidade Carmela Dutra, Rio de Janeiro, Rio de Janeiro
  - Hospital Maternidade Alexandre Fleming, Rio de Janeiro, Rio de Janeiro
  - Hospital Geral de Bonsucesso, Rio de Janeiro, Rio de Janeiro
  - Instituto Fernandes Figueira, Rio de Janeiro, Rio de Janeiro
  - Hospital Cachoeirinha, Cachoeirinha, Rio Grande do Sul
  - Hospital Femina, Porto Alegre, Rio Grande do Sul
  - Grupo Hospital Criança Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Alvorada, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Isabel, Aracaju, Sergipe
  - Maternidade Hildete Falcao Batista, Aracaju, Sergipe
  - Faculdade de Medicina de Botucatu - UNESP, Botucatu, São Paulo
  - Universidade de Campinas - UNICAMP, Campinas, São Paulo
  - HC da Fac. de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Matern. Escola de Vila Nova Cachoeirinha, São Paulo, São Paulo
  - Instituto da Criança - HCFMUSP, São Paulo, São Paulo
  - Hospital Universitario - USP, São Paulo, São Paulo

REFERENCES:
- [Background] Precioso AR, Sakae PP, Mascaretti RS, Kubrusly FS, Gebara VC, Iourtov D, Rebello CM, Vaz FA, Raw I. Analysis of the immunogenicity and stability of a porcine pulmonary surfactant preparation administered in rabbits. Clinics (Sao Paulo). 2006 Apr;61(2):153-60. doi: 10.1590/s1807-59322006000200011. Epub 2006 Apr 25. PMID 16680333
- [Background] Lyra JC, Mascaretti RS, Precioso AR, Haddad LB, Mauad T, Vaz FA, Rebello CM. Polyethylene glycol addition does not improve exogenous surfactant function in an experimental model of meconium aspiration syndrome. Exp Lung Res. 2009 Feb;35(1):76-88. doi: 10.1080/01902140802415837. PMID 19191106
- [Derived] Rebello CM, Precioso AR, Mascaretti RS; Grupo Colaborativo do Estudo Brasileiro Multicentrico de Surfactante. A multicenter, randomized, double-blind trial of a new porcine surfactant in premature infants with respiratory distress syndrome. Einstein (Sao Paulo). 2014 Oct-Dec;12(4):397-404. doi: 10.1590/S1679-45082014AO3095. PMID 25628188